CLINICAL TRIAL: NCT06187077
Title: Techquity by FAITH!: A Cluster Randomized Controlled Trial To Assess the Efficacy of a Community-informed, Cardiovascular Health Promotion Mobile Intervention With Digital Health Advocate Support
Brief Title: Techquity by FAITH!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Johns Hopkins University (Other); Association of Black Cardiologists (Unknown)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-011118; 3P50MD017342-03S3 (NIH)
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Health Equity; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA-Enhanced FAITH! App (Experimental): This group will use the FAITH! App with guided support from a Digital Health Advocate (DHA) within their church.
  Interventions: Behavioral: DHA-Enhanced FAITH! App
- FAITH! App (Other): This group will use the FAITH! App on their own, with no DHA support.
  Interventions: Behavioral: FAITH! App

INTERVENTIONS:
Behavioral: DHA-Enhanced FAITH! App — This group of participants will follow an 11-week guided intervention with the FAITH! App. Weekly educational modules provide information on components of cardiovascular health (CVH). Participants are given a Fitbit to track physical activity, which will automatically synch to the app and will be asked to track their daily fruit and vegetable intake on the app. DHAs will promote CVH and digital health readiness as peer mentors by guiding participants through the educational modules and encouraging use of the additional interactive app features. During the guided intervention phase, they will facilitate weekly visits with participants in their church, which will follow the FAITH! App modules and integrate a digital health topic. Following the 11-week guided intervention, participants will have a 12-month maintenance phase with access to use the app as they wish.
  Arms: DHA-Enhanced FAITH! App
Behavioral: FAITH! App — This group of participants will follow an 11-week guided intervention with the FAITH! App. Each week, an educational module is completed in the app, which provides information on a component of cardiovascular health. Participants will be given a Fitbit to track their physical activity, which will automatically synch to the app, and will be asked to track their daily fruit and vegetable intake on the app as well. Following the 11-week guided intervention, participants will have a 12-month maintenance phase in which they will have access to use the app as they wish.
  Arms: FAITH! App

SUMMARY:
The goal of this clinical trial is to engage African-American churches via an established community-academic partnership (FAITH! Program) to build capacity to promote cardiovascular health and digital health equity in African-American faith communities. There are 3 study aims:

Aim 1: Co-design a culturally tailored digital health equity toolkit with community members

Aim 2: Train a network of Digital Health Advocates (DHAs) in digital health equity and cardiovascular health promotion

Aim 3: Test the impact of a DHA-enhanced mobile health intervention (the FAITH! App) on cardiovascular health and digital health readiness among participants

In Aim 1, participants will attend a series of focus groups to share their input on a digital health equity curriculum that will be condensed into a toolkit.

In Aim 2, DHAs will be trained using this toolkit as well as a community health advocacy curriculum to learn how to promote digital health readiness and cardiovascular health in their communities.

Finally, Aim 3 will be a randomized controlled trial where participants will use the FAITH! App to improve their cardiovascular health. Some participants will have the added support of a DHA, and the control group participants will use the app with no additional support to test whether the DHA support is associated with a more significant improvement in cardiovascular health.

DETAILED DESCRIPTION:
This study addresses cardiovascular health and digital health disparities faced by African-Americans (AAs). We propose three aims to engage with the AA community and build capacity for a digital literacy and cardiovascular health promotion. Aim 1 will engage AA churches to co-design a culturally relevant digital health equity toolkit through an iterative focus group process. In aim 1, we will recruit 20 AAs to represent their churches and be trained as digital health advocates (DHAs) by completing digital health readiness education (using the toolkit developed in aim 1) and cardiovascular health promotion. This advocacy program will be integrated into an existing mobile health intervention, the FAITH! App, in Aim 3. The impact of the community-informed, mHealth intervention, enhanced with DHA support, on AA adults' cardiovascular health will be assessed in a cluster randomized controlled trial. 150 participants will be be randomized to utilize the FAITH! App alone or with the support of the DHA at their church. Cardiovascular health will be assessed at baseline, approximately 3 months, 6 months, and 12 months post-randomization using the American Heart Association's Life's Essential 8 metric for cardiovascular health.

ELIGIBILITY:
Aim 1- Inclusion Criteria: African/American race/ethnicity, age ≥ 18 years, basic Internet navigation skills, active email address

Aim 2- Inclusion Criteria: African/American race/ethnicity, age ≥ 18 years, ownership of smartphone (supporting iOS or Android systems), moderate to high digital health literacy (by eHealth literacy scale [eHEALS], score ≥26)

Aim 3- Inclusion Criteria: African/American race/ethnicity, age ≥ 18 years, ownership of smartphone (supporting iOS or Android systems), low digital health literacy (by eHEALS, score ≤26), basic Internet navigation skills, at least weekly Internet access, active email address, fruit/vegetable intake ≤5 servings/day, no regular physical activity, able to engage in moderate physical activity and willingness to participate in all aspects of the study.

Exclusion Criteria: Unable to walk up ≥2 flights of stairs or walk ≥1 city block without assistance or stopping, pregnant (at time of study enrollment), visual/hearing impairment or mental disability that would preclude independent app use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Life's Essential 8 Composite Score change | Baseline, 6-months and 12-months post-randomization
  Changes from baseline in Life's Essential 8 score. Life's Essential 8 composite score is determined as a composite of all components by calculating an unweighted average score on a scale of 0 to 100 points. An overall cardiovascular health score (Life's Essential 8 score) will be considered high (80 to 100 points), moderate (50 to 79 points) or low for (0 to 49 points).
Blood Pressure Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Average of 3 sitting measurements of systolic and diastolic pressures (mmHg).
Fasting Glucose/Hemoglobin A1c Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Fingerstick blood collection (fasting glucose-mg/dL; Hemoglobin A1c-%).
Fasting Blood Lipids Score Change (non-HDL cholesterol) (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Fingerstick blood collection (mg/dL).
Body Mass Index (BMI) Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Calculated by weight (kg) and height (m).
Tobacco/Nicotine Exposure Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Changes from baseline in smoking status using the National Health and Nutrition Examination Survey-Smoking-Cigarette Use Questionnaire (NHANES-SMQ), evaluating current and past tobacco use habits.
Dietary Quality Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Changes from baseline in healthy diet using the Mediterranean Eating Patterns for Americans (MEPA), a 16-item questionnaire evaluating accordance with a Mediterranean-like diet pattern.
Physical Activity Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Change from baseline in the total minutes per week that a participant engaged in moderate and vigorous intensity physical activity at immediate post-intervention. Physical activity will be measured by the International Physical Activity Questionnaire (IPAQ).
Sleep Health Score Change (Life's Essential 8 Component) | Baseline, 6-months and 12-months post-randomization
  Changes from baseline in sleep quality (number of hours of sleep nightly) using the Pittsburg Sleep Quality Index (PSQI).

SECONDARY OUTCOMES:
Digital Health Readiness | Baseline, 3 months post-randomization
  Assessed using a validated, 20-item instrument that captures 5 domains: digital skills, digital usage, digital literacy, digital health literacy, and digital learnability adapted for all digital health technologies such as smartphone apps.
Social Support - Diet | Baseline, 3 months, 6 months, and 12 months post-randomization
  Diet social support measured using the Social Support for Eating Habits Survey scale. This scale assesses the level of encouragement or discouragement from family and friends that participants received for adopting healthier eating habits. 5 questions were asked to assess the degree of encouragement and discouragement, separately, on a 5-point scale [from 1 (none) to 5 (very often)]. Each sub-item was summed to obtain a score ranging from 5 (lowest) to 25 (highest discouragement/encouragement). The change in level of diet social support was calculated from baseline to 6 months post-intervention. Higher scores indicate more change in social support for healthy eating.
Self Regulation - Diet | Baseline, 3 months, 6 months, and 12 months post-randomization
  Diet self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to eat healthier foods. Items are measured on a five-point scale from 1 (never) to 5 (always). A mean of all items is obtained and a difference between the scores is calculated. Higher change in scores indicate more change in use of self-regulation strategies to promote healthy eating.
Perceived Barriers - Diet | Baseline, 3 months, 6 months, and 12 months post-randomization
  Changes from baseline to 12 months post-intervention in diet perceived barriers measured by Barriers to Diet and Exercise questionnaire. The 39-item instrument is measured on a five-point scale from 1 (not at all true for me) to 5 (very true for me); participants indicate the extent to which each factor has made it difficult for them to follow appropriate eating and exercise habits in the past 6 months.
Social Support - Physical Activity | Baseline, 3 months, 6 months, and 12 months post-randomization
  Physical activity social support measured using the Social Support for Exercise Survey scale. This scale assesses the level of encouragement or discouragement from family and friends that participants received for adopting healthier physical activity habits. 5 questions were asked to assess the degree of encouragement and discouragement, separately, on a 5-point scale [from 1 (none) to 5 (very often)]. Each sub-item was summed to obtain a score ranging from 5 (lowest) to 25 (highest discouragement/encouragement). The change in level of physical activity social support was calculated from baseline to 6 months post-intervention. Higher scores indicate more change in social support for physical activity. Family Participation was calculated as a sum of 10 items: 10 = low to 50 = high; Family Rewards/Punishment as a sum of 3 items: 3 = low to 15 = high; and Friend Participation sum of 10 items: 10 = low to 50 = high.
Self Regulation - Physical Activity | Baseline, 3 months, 6 months, and 12 months post-randomization
  Physical activity self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to increase their step count or physical activity levels. Items are measured on a 10-item five-point scale from 1 (never) to 5 (always). The mean of the ten items is obtained. The difference in the mean scores from baseline to 6 months post-intervention is calculated. Larger change in scores indicate more change in self-regulation.
Perceived Barriers - Physical Activity | Baseline, 3 months, 6 months, and 12 months post-randomization
  Changes from baseline to 12 months post-intervention in diet perceived barriers measured by Barriers to Diet and Exercise questionnaire. The 39-item instrument is measured on a five-point scale from 1 (not at all true for me) to 5 (very true for me); participants indicate the extent to which each factor has made it difficult for them to follow appropriate eating and exercise habits in the past 6 months.
Artificial Intelligence (AI)-Electrocardiogram (ECG) | Baseline, 6 months and 12 months post-randomization
  Standard 12-lead ECG to be analyzed by a Mayo Clinic AI-enhanced ECG model for detection of left ventricular dysfunction and correlation of actual age and AI-ECG predicted age.
Cardio-ankle vascular index (CAVI) | Baseline, 6 months and 12 months post-randomization
  The cardio-ankle vascular index (CAVI) is a measure of arterial stiffness that reflects the stiffness from the ascending aorta to the ankle arteries. Normal CAVI values are less than 8 and values greater than or equal to 9 are classified as abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess Brewer, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT06187077/ICF_000.pdf